CLINICAL TRIAL: NCT06365229
Title: Percutaneous Unilateral Biportal Endoscopy Versus Uniportal Endoscopy for Lumbar Spinal Stenosis: a Single-center, Prospective, Non-randomized Cohort Trial Protocol
Brief Title: Percutaneous Unilateral Biportal Endoscopy Versus Uniportal Endoscopy for Lumbar Spinal Stenosis: Study Protocol
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-P2-336-02
Record Dates: First submitted 2024-04-07; First posted 2024-04-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- UBE Group: Patients with LSS undergoing UBE
- UE Group: Patients with LSS undergoing UE

SUMMARY:
A prospective study aimed to compare the efficacy and safety of Unilateral biportal endoscopic (UBE) technique and uniportal endoscopic (UE) technique for treating patients with lumbar spinal stenosis (LSS).

ELIGIBILITY:
Inclusion Criteria:

* Age range: 50-80 years
* Diagnosed with LSS of 1-2 response levels
* The predominant manifestation is neurogenic intermittent claudication, and conservative treatment has been ineffective for at least 3 months
* Degenerative lumbar spondylolisthesis of less than I degree or without spine instability
* Patients agree to participate in the study and are willing to complete the follow-up

Exclusion Criteria:

* Isthmic lumbar spondylolisthesis or degenerative lumbar spondylolisthesis of greater than I degree
* Instability at the response level
* Prior surgical history at the response level
* Scoliosis with Cobb angle >20 degrees
* Other conditions affecting the lumbar spine (infection, tumor, fracture, neurological diseases, and others)
* Patients with medical disorders who are unable to tolerate surgery

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with LSS undergoing UBE or UE decompression performed by two experienced spine surgeons at the same hospital will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | From enrollment to the end of follow-up at 1 year
  0-100%, the higher the score, the more severe the lumbar spine dysfunction

SECONDARY OUTCOMES:
Magnetic resonance imaging (MRI) | From enrollment to the follow-up at 2 weeks
  Enlargement ratio of the dural sac
Computed tomography (CT) scans | From enrollment to the end of follow-up at 2 weeks
  bony decompression range; preservation rate of the facet joint
Creatine kinase (CK) | From enrollment to the end of follow-up at 2 weeks
Erythrocyte sedimentation rate (ESR) | From enrollment to the follow-up at 2 weeks
Surgical complication | From enrollment to the end of follow-up at 1 year
  Adverse events will be recorded to assess the safety of decompression using UBE or UE for LSS.
VAS (visual analogue scale) for leg pain | From enrollment to the end of follow-up at 1 year
  0-10, the higher the score, the more severe the pain
VAS (visual analogue scale) for lower back pain | From enrollment to the end of follow-up at 1 year
  0-10, the higher the score, the more severe the pain
Japanese Orthopaedic Association (JOA) score | From enrollment to the end of follow-up at 1 year
  0-29, the higher the score, the better the lumbar spine function
Modified MacNab criteria | From enrollment to the end of follow-up at 1 year
  According to satisfaction, it is divided into four levels: excellent, good, acceptable, and poorexcellent, good, fair, and poor
Operation time | Immediately after the surgery
Blood loss | Immediately after the surgery
Postoperative hospital stays | Immediately after the discharge
Age | Baseline, pre-surgery
Gender | Baseline, pre-surgery
Body mass index (BMI) | Baseline, pre-surgery
Medical comorbidity | Baseline, pre-surgery
Smoking status | Baseline, pre-surgery
Alcohol status | Baseline, pre-surgery
Symptoms duration | Baseline, pre-surgery
Physical examination finding | Baseline, pre-surgery
Previous spinal surgery | Baseline, pre-surgery
Affected level | Baseline, pre-surgery
Stenosis grade | Baseline, pre-surgery
Physical-component summary score of the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | From enrollment to the end of follow-up at 1 year
  range, 0-100 points, with higher scores indicating better physical health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan H, Liu Y, Li G, Yu L, Yang Y, Lo Y, Bin Z, Li X. Percutaneous unilateral biportal endoscopy versus uniportal endoscopy for lumbar spinal stenosis: a single-centre, prospective, non-randomised cohort trial protocol. BMJ Open. 2025 Jul 25;15(7):e087863. doi: 10.1136/bmjopen-2024-087863. PMID 40713043